CLINICAL TRIAL: NCT00133601
Title: Cognitive Behavioral Therapy for Insomnia in Chronic Pain Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Michael Perlis; Associate Professor, Psychiatry; Director, Behavioral Sleep Medicine Program, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9080; 5R21NR009080-02 (NIH)
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Insomnia; Chronic Pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CBT-1
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT-I including sleep restriction, stimulus control, sleep hygiene instructions and one session of cognitive therapy devoted to catastrophic thoughts about the consequences of insomnia.
  Arms: 1

SUMMARY:
This study of cognitive behavioral therapy for insomnia in chronic pain patients is a randomized, controlled clinical trial of parallel groups with three and six months follow up.

DETAILED DESCRIPTION:
Forty five subjects, both male and female, of diverse racial backgrounds, ages >25 with insomnia secondary to pain will be recruited from the Pain Clinic at URMC and from the community at large via advertisements and solicited primary care referrals to participate in a parallel-groups, randomized, single blind, controlled trial. Protocol eligible subjects (as determined via a phone screen interview or by responses to our web based screening questionnaire) will be evaluated in-lab. The screen will determine whether subjects have chronic insomnia secondary to pain and do not meet any of the exclusion criteria. Once found to be study eligible, they are given an appointment for the reading and signing of the consent and the intake interview. The in-lab intake interview includes the administration of a broad battery of self-report instruments. Following the clinical interview, subjects will undergo a physical exam. The history (to include drug and ETOH use) and physical examination will include blood and urine chemistries to rule out any acute or unstable medical co-morbidity (including pregnancy). The lab work will include profiles to assess renal, liver, thyroid, and anemia as well as urine toxicology screen for illicit drug use. The lab work results will be reviewed by the Co-PI and our medical consultant. If significant abnormal findings are discovered, the subject will be referred to their primary care provider for treatment. In addition to conducting an "in-house" physical, after the subject signs a release of information, the researchers also FAX the prospective subject's primary care physician a letter asking them to confirm that the individual is eligible for the study.

If data from both these evaluations suggest that the subject is protocol eligible, according to the inclusion and exclusion criteria, the subject is asked to fill out two weeks of sleep/pain diaries. The diary data are used to "prospectively" confirm the severity and frequency of the subjects sleep complaints and as baseline data. Finally, all subjects will be evaluated by polysomnography (PSG) to assure that they do not have an occult sleep disorder. Once determined to be study appropriate, the subjects will be randomized into a treatment group. They will see the therapist weekly for 8 weeks. At 3 month and 6 month intervals after weekly therapy session end, the subject will be asked to fill out sleep diaries and wear an actiwatch for a period of two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for Study: Over 25 years of age
* Chronic pain (>6 months) in the neck and back that has been diagnosed by a physician
* Insomnia (>30 minutes to get to sleep, >30 minutes wake during the night and daytime loss of function due to insomnia and pain)

Exclusion Criteria:

* Unstable medical problems
* Currently undergoing surgery or procedures for their pain or medical problems
* Head injuries
* Seizure disorders
* Taking sleeping pills

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-10; Primary Completion 2007-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine and confirm "prospectively" the severity and frequency of the subjects sleep complaints and as baseline data. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perlis, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Neurophysiology and Sleep Research Laboratory, Rochester, New York, United States